CLINICAL TRIAL: NCT06895122
Title: Effectiveness of High-speed Resistance and Multicomponent Training in Older Adults With Sarcopenic Obesity: a Randomized Clinical Trial
Brief Title: Effectiveness of Different Types of Training in Older Adults With Sarcopenic Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Luis Polo Ferrero, Associate Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OB_SARC_
Record Dates: First submitted 2025-03-18; First posted 2025-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Sarcopenic Obesity; Obesity and Overweight; Sarcopenia
Keywords: Resistance training; Exercise; Older adults; Multicomponent training
MeSH Terms: conditions — Obesity; Overweight; Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Longitudinal.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding was performed on the study hypothesis and on the participants assigned to each group. Both the evaluating researchers and the statistical researcher were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Speed Resistance Training (Experimental): The core component of the H-RT program will include a variety of exercises targeting both the upper and lower limbs. These exercises consist of wall push-ups, arm raises, elbow flexion and extension, weighted pronosupination, hand presses, knee and hip hinge squats, deadlifts, frontal and sagittal plane lunges, and heel raises. The program will be structured into three progressive phases:
  Phase 1 - Adaptation: During the first month, participants will focus on learning the correct technique for all upper and lower limb exercises to ensure proper execution.
  Phase 2 - Strength Training: Over the next two months, resistance exercises will be performed at both slow and controlled speeds, reinforcing movement patterns established in the initial phase.
  Phase 3 - High-Speed Resistance Training: In the final five months, progressive overload will be applied, with a gradual increase in execution speed and exercise intensity to enhance muscle power and improve overall function
  Interventions: Procedure: High resistance training
- Multicomponent training (Active Comparator): The core of the multicomponent exercise program incorporates various exercise modalities, including aerobic training, mobility, strength, balance, and coordination exercises. Additionally, playful activities and cognitive tasks are integrated to enhance the program's overall effects. These include games involving colors, numbers, letters, laterality (right-left distinction), memory exercises, and more. The progression for each modality follows a structured approach:
  Aerobic Training: Begins with continuous exercise, transitions to interval training, and progressively reduces rest periods.
  Strength Training: Gradually increases the number of sets and repetitions while decreasing rest time.
  Balance Training: Starts with static exercises and progresses to more challenging tasks, incorporating blindfolds, perturbations, and dynamic balance drills.
  Coordination and Cognitive Tasks: Exercises become progressively more complex, requiring faster decision-making and more intricate movements.
  Interventions: Procedure: Multicomponent Training
- Control Group (No Intervention): Participants assigned to this group will maintain their usual dietary habits and physical activity levels without making any lifestyle modifications throughout the study. They will not engage in the muscle power-based strength training program or participate in any other structured, supervised, or systematic exercise program.

INTERVENTIONS:
Procedure: High resistance training — Participants will perform the exercises at high speed, emphasizing explosive movements to maximize muscle power development.
  Other Names: Power training
  Arms: High Speed Resistance Training
Procedure: Multicomponent Training — Various exercise modalities are integrated, including aerobic training, mobility, strength, balance, and coordination exercises.
  Arms: Multicomponent training

SUMMARY:
This study is a randomized, parallel-group, double-blind clinical trial. The primary aim is to assess the effectiveness of power-based resistance training, multimodal exercise incorporating non-specific movements, and a control group in improving functionality and body composition in women over 65 years old with pre-sarcopenia. The intervention will take place over 30 weeks, with three training sessions per week in both experimental groups. Assessments will be conducted at two time points: before and after the intervention. Evaluated parameters will include functionality (Timed Up & Go test (TUG), chair stand test, handgrip strength, and Short Physical Performance Battery (SPPB)) and body composition (body fat percentage, skeletal muscle index (SMI), appendicular skeletal muscle mass (ASM), waist circumference, waist-to-hip ratio, body weight, and body mass index (BMI)).

DETAILED DESCRIPTION:
Design: This study is a randomized controlled clinical trial with three parallel groups, recruiting women over 65 years old with sarcopenic obesity. Participants will be randomly assigned to one of three intervention groups. The study will span 8 months, with two assessment points: an initial evaluation and a final follow-up at 8 months. Throughout the intervention period, participants will attend three supervised sessions per week, each lasting 50 minutes.

Setting: The study will take place in the Salamanca Health Area, in collaboration with the Research, Teaching, and Care Unit of the Faculty of Nursing and Physiotherapy at the University of Salamanca and the Department of Older Adults of the Salamanca City Council.

Interventions: The three intervention groups include: (1) a Multicomponent Exercise Program (MT); (2) a Muscle Strength Training Program (M-RT); and (3) a Control Group (CG) with no structured exercise intervention. Both MT and M-RT sessions will follow a standardized format, incorporating exercises based on the guidelines of the American College of Sports Medicine (ACSM). The strength component of the MT program will progressively increase in speed, adjusting to the maximum capability of each participant.

Study Population: A total of 33 women aged 65 years and older with sarcopenic obesity, residing in Salamanca, will be enrolled and randomly allocated into the three study groups in a 1:1:1 ratio. Randomization will be carried out using Epidat 4.2 software, and the sample size was determined using GRANMO version 8.

Outcome Measures: The primary outcome is the Skeletal Muscle Index (SMI). Secondary outcomes include functional assessments (Timed Up & Go [TUG] test, chair rise test, handgrip strength test, and Short Physical Performance Battery [SPPB]), body composition measures (percentage of body fat, appendicular skeletal muscle mass [ASM], waist circumference, waist-to-hip ratio, body weight, and body mass index [BMI]), and gait speed. Descriptive statistics will be reported as mean ± standard deviation for continuous variables and as frequency distributions for categorical variables.

Statistical Analysis: Normality tests and baseline comparisons will be conducted to confirm group homogeneity. Depending on data distribution, parametric or non-parametric tests will be applied to assess intra-group changes. To compare the effects between groups, repeated measures ANOVA will be used when assumptions of normality and sphericity are met, whereas mixed-effects models will be applied for handling missing data. If normality is violated, the Kruskal-Wallis test will be used. When significant differences are found, post-hoc comparisons will be performed using Bonferroni or Tukey corrections. A significance level of α = 0.05 will be considered. All statistical analyses will be conducted using SPSS version 28.0.

Ethical Considerations: The study has received approval from the Ethics Committee for Drug Research (CEIm) of the Salamanca Health Area. All participants will provide informed consent after being fully briefed on the study's objectives, potential risks, and expected benefits. The research follows the ethical principles outlined in the Declaration of Helsinki, Law 14/2007 on Biomedical Research, and other relevant legal and ethical guidelines applicable to the study's nature.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 65 years.
* Diagnosis of sarcopenic obesity (SMI < 5.5 kg/m2, BMI > 30 kg/m2)

Exclusion Criteria:

* Tumors
* Pacemakers
* Fibrillations
* Cardiac pathology or uncontrolled hypertension
* History of severe trauma/recent cervical surgery
* Uncontrolled systemic and inflammatory pathologies
* Congenital collagen compromise
* Presence of difficulties in performing the Initial Evaluation tests
* Language barriers
* Pending litigation or legal claim

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Only individuals who self-identify as women and meet the biological criteria of the study (i.e., assigned female at birth) are eligible to participate
Enrollment: 33 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Index (SMI) | 30 weeks
  The SMI assesses muscle mass relative to body size, calculated as appendicular skeletal muscle mass (ASM) divided by height squared (kg/m²). Sarcopenia is diagnosed in women when SMI is <5.5 kg/m²

SECONDARY OUTCOMES:
Body Fat Percentage (BF%) | 30 weeks
  BF% represents the proportion of total body weight composed of fat mass. It is a key indicator of body composition and metabolic health, with higher values often associated with increased health risks.
Grip strength test | 30 weeks
  Accurate measurement of hand grip strength requires the use of a hand dynamometer (Jamar Plus) calibrated under well-defined (standardized) test conditions. Force values less than 16 Kg are considered positive.
Chair stand test | 30 weeks
  It can be used as an indicator of the strength of the lower limb muscles. It measures the amount of time a patient needs to get up five times from a sitting position without using their arms. It will help us to affirm that the person has a probable sarcopenia. Times greater than 15 seconds are considered positive
Body Mass Index (BMI) | 30 weeks
  BMI is a measure used to assess body weight in relation to height, calculated as weight in kilograms divided by height in meters squared (BMI = kg/m²). A BMI of 30 kg/m² or higher is classified as obesity.
Short Physical Performance Battery (SPPB) | 30 weeks
  Test to assess physical performance and degree of frailty consisting of 3 subtests: gait speed, balance, and lower limb strength. The maximum score is 12 points and a score ≤ 8 points indicates poor physical performance.
Gait speed | 30 weeks
  It is considered a fast, safe and very reliable test for sarcopenia, in a distance of 4 meters, values greater than 0.8 m/s are considered positive.
Timed Up and Go (TUG) | 30 weeks
  A predictive test for frailty and falls, where individuals are asked to get up from a standard chair, walk to a marker 3 m away, turn around, and sit down again. Times greater than 20 seconds are considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Méndez Sánchez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- University of Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided